



'Implementation and Validation of the Dutch Translation of the TAPS-tool: a Screener for Tobacco, Alcohol, Prescription Medication and Other Substances for Patients With Severe Mental Illness With and Without Intellectual Disabilities'

ECSW-2021-052

Date 19.04.2021





**Date** 19 april 2021

Subject Participation on research on the TAPS-tool

Dear sir / madame,

Because of your treatment within ORO, you will shortly be asked to complete a questionnaire about substance use (smoking, alcohol, drugs), this is the SumID-Q.

#### Something new:

A number of practitioners within the GGZ Oost Brabant are preparing a new questionnaire about substance use that is shorter than the questionnaire you are currently receiving. This new questionnaire is called the TAPS. We think it is important that we have a short questionnaire so that we know from as many people as possible whether there is substance use. This is important to be able to give everyone good treatment.

# Research:

Before we can use this new questionnaire (the TAPS), we must first investigate whether this is a good questionnaire. We ask for your cooperation for this investigation. Your cooperation is voluntary, but we do need your written consent.

### If you participate:

If you participate, in addition to the SumID-Q, for which you have an appointment, the TAPS will also be administered once by the practitioner or nurse. These are some additional questions about smoking, drugs, alcohol and medicines. Those extra questions will take a maximum of half an hour. You decide whether you want to participate. If you do not participate, this will not affect your treatment.

If you do participate, you can always change your mind and indicate that you no longer want to participate. You don't have to say why you're stopping. We will then not use your data for the research.

#### What will happen to your answers:

We want to save your answers to the 2 questionnaires, the SumID-Q and the TAPS in a computer file in the secure environment of the GGZ. We would also like to add a few other details such as your gender, age and diagnosis. To protect your privacy, your data is given a code. This is called anonymous processing of the data. Your name, and other information that may identify you as a person, will be omitted and replaced by this code. The data can only be traced back to you with the key of the code. This key is safely stored within the ORO foundation. Only the data with the

code will be passed on to the GGZ. In order to ultimately be able to say how good the TAPS questionnaire is, only the codes are used. Even when we write down the results of this research in a report, only the anonymous data is used and statements are made about the entire group of people who participated in this research.

The answers and your other data are entered by the researchers, who look in your file for this. Your answers to the TAPS questionnaire must be kept for 15 years.

#### Informed consent form:

If you give permission, we will ask you to confirm this in writing on the corresponding declaration of consent. By your written consent, you indicate that you have understood the information and agree to participate in the study. Both you and the researcher will receive a signed version of this consent form.

Would you like to know more? Then you can call Birgit Seelen (telephone: 06-81405847).

Kind regards,

Birgit Seelen, GZ psychologist / researcher

## CONSENT FORM: Research into the TAPS questionnaire

I want to participate tot his research:

- I've read the information letter. I could also ask questions. My questions have been sufficiently answered. I had plenty of time to decide whether to participate.
- I know that taking part is voluntary. I also know that I can decide at any time not to participate or to stop the study. I don't have to give a reason for that.
- I give permission for the collection and use of my answers to answer the research question in this study.
- I know that the researchers need my answers and some other data for this. I give the researchers permission to use this data.

| Name of subject:<br>Signature: | Date | :_/_/_ |
|---|---|---|
| Name mentor/curator (if applicable): Signatur: | Date | :_/_/_ |
| I declare that I have fully informed this subject about the said | study. | |
| Name investigator (or representative): Signature: | Date: _ | _/_/_ |

The subject receives a complete information letter, together with a signed version of the consent form



